CLINICAL TRIAL: NCT00466817
Title: A Phase III, Randomized, Placebo-Controlled Blinded Investigation of Six Weeks vs. Six Months of Oral Valganciclovir Therapy in Infants With Symptomatic Congenital Cytomegalovirus Infection (CASG 112)
Brief Title: Short-Term vs. Long-Term Valganciclovir Therapy for Symptomatic Congenital CMV Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-0046; CASG 112
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Cytomegalovirus Infection
Keywords: Cytomegalovirus, congenital, infants
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Valganciclovir (Experimental): Six months of oral Valganciclovir.
  Interventions: Drug: Valganciclovir
- Placebo (Placebo Comparator): Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
  Arms: Placebo
Drug: Valganciclovir — Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
  Arms: Valganciclovir

SUMMARY:
Cytomegalovirus (CMV) infection is known to cause hearing loss and mental retardation. The purpose of this study is to compare a 6-week course to a 6-month course of the drug valganciclovir in babies born with CMV to assess the safety and efficacy of this treatment. Participants will include 104 infants (30 days old or younger) born with CMV disease. All infants will take valganciclovir by mouth for 6 weeks. At the end of the 6 week period, subjects will be assigned by chance to receive either valganciclovir or placebo (inactive substance) to complete the 6 months of antiviral treatment. Patients will be followed for the study related evaluations of safety, changes to hearing, and developmental milestones for up to 2 years. Patients will be followed by telephone contact for an additional 3 years. Thus, participants may be involved in study related procedures for approximately 5 years.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, international, Phase III, randomized and blinded investigation of 6 weeks versus 6 months of oral valganciclovir therapy in babies with symptomatic congenital cytomegalovirus (CMV) disease. Following enrollment, study subjects will receive 6 weeks of oral valganciclovir. Near the end of the 6-week course, subjects will be randomized in a 1:1 fashion either to continue on valganciclovir to complete 6 months of therapy or to begin a matching placebo to complete the 6 months. Study subjects will be stratified according to whether or not there is central nervous system (CNS) involvement at study entry. During the 6-month treatment period and the 1 month thereafter, study subjects will be followed weekly for 4 weeks, then every other week for 8 weeks, then every month for 4 months. At each of these visits, safety labs will be checked, growth parameters recorded, and adverse events assessed. The dose of study medication will be adjusted for weight gain at each of these study visits. Dose adjustments may also occur as indicated per protocol for neutropenia, thrombocytopenia, or renal impairment. Whole blood will be obtained for CMV viral load at each of these visits as well. Hearing outcomes will be assessed at baseline, 6 months, 12 months and 24 months. Developmental outcomes will be assessed at 12 months and 24 months. Changes in whole blood viral load measurements will be correlated with both hearing and neurologic outcomes. In study subjects with increasing whole blood viral loads during the course of treatment, assessment for antiviral resistance may be undertaken.Safety assessments include: hematology labs, chemistry labs, physical examinations, and adverse event data performed/collected serially. Development of neutropenia will be confirmed by repeat blood testing within one week, and study drug will be held until it resolves. Efficacy assessments include: hearing assessments at baseline, 6 months, 12 months and 24 months; and neurodevelopmental assessments at 12 months and 24 months. Study objectives are: to compare the impact on hearing outcomes of 6 weeks versus 6 months of antiviral treatment with valganciclovir oral solution in infants with symptomatic congenital CMV disease; to compare the safety profile of 6 weeks versus 6 months of antiviral therapy with valganciclovir oral solution in infants with symptomatic congenital CMV disease; to compare the impact on neurologic outcomes of 6 weeks versus 6 months of antiviral treatment with valganciclovir oral solution in infants with symptomatic congenital CMV disease; and to correlate change in whole blood viral load with hearing and neurologic outcomes. Participants will include 104 male and female neonates (less than or equal to 30 days) with symptomatic congenital CMV.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s)
* Confirmation of cytomegalovirus (CMV) from urine or throat swab specimens by culture, shell vial, or polymerase chain reaction (PCR) tests
* Symptomatic congenital CMV disease, as manifest by one or more of the following:

  1. Thrombocytopenia
  2. Petechiae
  3. Hepatomegaly
  4. Splenomegaly
  5. Intrauterine growth restriction
  6. Hepatitis (elevated transaminases and/or bilirubin)
  7. Central nervous system (CNS) involvement of the CMV disease [such as microcephaly, radiographic abnormalities indicative of CMV CNS disease, abnormal cerebrospinal fluid (CSF) indices for age, chorioretinitis, hearing deficits as detected by formal brainstem evoked response (not a screening auditory brainstem response {ABR}), and/or positive CMV PCR from CSF]
* Less than or equal to 30 days of age at study enrollment
* Weight at study enrollment greater than or equal to 1800 grams
* Gestational age greater than or equal to 32 weeks at birth

Exclusion Criteria:

* Imminent demise
* Patients receiving other antiviral agents or immune globulin
* Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., a history of necrotizing enterocolitis)
* Documented renal insufficiency, as noted by a creatinine clearance less than 10 mL/min/1.73m^2 at time of study enrollment
* Breastfeeding from mother who is receiving ganciclovir, valganciclovir, foscarnet, cidofovir, or maribivir
* Infants known to be born to women who are human immunodeficiency virus (HIV) positive (but HIV testing is not required for study entry)
* Current receipt of other investigational drugs

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (41):
  - University of Alabama - Children's of Alabama - Clinical Virology, Birmingham, Alabama
  - University of South Alabama - Children's Specialty Clinic, Mobile, Alabama
  - Arkansas Children's Hospital - Infectious Diseases, Little Rock, Arkansas
  - Los Angeles County - University of Southern California - Medical Center - Pediatrics, Los Angeles, California
  - Plaza Towers Obstetrics and Gynecology, Los Angeles, California
  - Children's Hospital of Orange County - Infectious Diseases, Orange, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado - Infectious Disease, Aurora, Colorado
  - Children's National Medical Center - Sheikh Zayed Campus - Infectious Disease, Washington D.C., District of Columbia
  - University of Florida - College of Medicine - Jacksonville, Jacksonville, Florida
  - University of South Florida - Tampa General Hospital - Pediatrics, Tampa, Florida
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Louisville School of Medicine - Kosair Childrens Hospital - Infectious Diseases, Louisville, Kentucky
  - Tulane University - Tulane Medical Center - Pediatrics, New Orleans, Louisiana
  - Louisiana State University Health Shreveport - Pediatrics, Shreveport, Louisiana
  - Johns Hopkins Children's Center - Pediatric Infectious Diseases, Baltimore, Maryland
  - Children's Hospital Boston - Infectious Diseases, Boston, Massachusetts
  - University of Minnesota - Pediatric Infectious Disease, Minneapolis, Minnesota
  - University of Mississippi - Children's Infectious Diseases, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - Creighton University Medical Center - Medicine - Infectious Diseases, Omaha, Nebraska
  - Childrens Hospital at Saint Peters University Hospital - Allergy, Immunology and Infectious Diseases, New Brunswick, New Jersey
  - Robert Wood Johnson Medical School - Pediatrics, New Brunswick, New Jersey
  - Women & Children's Hospital of Buffalo - Infectious Diseases, Buffalo, New York
  - Cohen Children's Medical Center - Pediatric Infectious Diseases, Manhasset, New York
  - University of Rochester Medical Center - Golisano Children's Hospital - Infectious Diseases, Rochester, New York
  - SUNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Carolinas Medical Center - Pediatrics - Infectious Diseases, Charlotte, North Carolina
  - MetroHealth Medical Center - Pediatric Infectious Disease, Cleveland, Ohio
  - Cleveland Clinic Main Campus - Center for Pediatric Infectious Diseases, Cleveland, Ohio
  - Nationwide Children's Hospital - Infectious Diseases, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC - Pediatric Infectious Diseases, Pittsburgh, Pennsylvania
  - Rhode Island Hospital - Pediatrics, Providence, Rhode Island
  - Medical University of South Carolina - Pediatrics - Infectious Diseases, Charleston, South Carolina
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee
  - Children's Medical Center Dallas - Neonatal ICU, Dallas, Texas
  - University of Texas Southwestern Medical Center - Pediatrics, Dallas, Texas
  - Cook Children's Infectious Disease Services, Fort Worth, Texas
  - University of Utah - Pediatric Pharmacology Program, Salt Lake City, Utah
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham, Birmingham
  - Bristol Royal Hospital for Children - UBHT Education Centre, Bristol, Bristol, City of
  - Alder Hey Childrens Hospital, Liverpool, Liverpool
  - University College London - Royal Free Campus - Virology, London, London, City of
  - Saint George's Hospital - Pediatric Infectious Diseases, London, London, City of
  - Newcastle General Hospital, Newcastle upon Tyne, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford, Oxfordshire

REFERENCES:
- [Derived] Kimberlin DW, Jester PM, Sanchez PJ, Ahmed A, Arav-Boger R, Michaels MG, Ashouri N, Englund JA, Estrada B, Jacobs RF, Romero JR, Sood SK, Whitworth MS, Abzug MJ, Caserta MT, Fowler S, Lujan-Zilbermann J, Storch GA, DeBiasi RL, Han JY, Palmer A, Weiner LB, Bocchini JA, Dennehy PH, Finn A, Griffiths PD, Luck S, Gutierrez K, Halasa N, Homans J, Shane AL, Sharland M, Simonsen K, Vanchiere JA, Woods CR, Sabo DL, Aban I, Kuo H, James SH, Prichard MN, Griffin J, Giles D, Acosta EP, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Valganciclovir for symptomatic congenital cytomegalovirus disease. N Engl J Med. 2015 Mar 5;372(10):933-43. doi: 10.1056/NEJMoa1404599. PMID 25738669

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 109 subjects started on valganciclovir. At the end of 6 weeks, subjects were randomized to valganciclovir or placebo. of the 109 subject that started, 12 dropped out before randomization and 1 subject was randomized but never received any blinded study drug.
Groups:
- Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo: Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
- Valganciclovir: 24 Wks of Valganciclovir: Six months of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
Period: Overall Study
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Started | 49 | 47
Completed | 44 | 43
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo: Six weeks of oral Valganciclovir followed by placebo (18 weeks) to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
- Valganciclovir: 24 Wks of Valganciclovir: Six months (6 weeks open label, 18 weeks blinded) of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
- Total: Total of all reporting groups
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir | Total
Number analyzed (Participants) | 49 | 47 | 96
Age, Continuous [Median (Full Range); unit: weeks] | 19 [2 to 30] | 14 [5 to 30] | 15 [2 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 29 | 31 | 60
Region of Enrollment [Number; unit: participants]
  United States | 49 | 47 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Ear Hearing Assessments at 6 Months.
Description: Hearing assessment was evaluated by an independent audiologist. At baseline, a brainstem evoked response (BSER) assessment and autoacoustic emissions (OAEs) hearing assessments were obtained. At 6 months, BSER and /or Visual reinforcement audiometry (VRA) and OAEs were obtained. A single, independent study audiologist who was blinded to treatment assignment assessed the audiology test battery for each subject and assigned the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications were assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. Following this, the study audiologist assigned the "best ear" classification for the subject at that study visit; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification was mild hearing loss.
Time Frame: Between baseline and 6 months
Population: Only subjects randomized and subjects that had both baseline and 6 month hearing exams were analyzed for the primary endpoint. Some subjects failed to have the one or both of the two hearing exams (baseline and/or 6 months). There were 43 subject in each group (placebo and active) that had both hearing results reported
Measure: Number; unit: participants
Groups:
- Placebo: 6 Wks Valganciclovir Followed by 18 Wks Placebo: Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 43 | 43
participants
  Worsened | 3 | 5
  No Change | 37 | 36
  One point improvement | 3 | 2

2. Secondary Outcome: Adverse Events Which Lead to Permanent Discontinuation of Valganciclovir Therapy or Lead to Irreversible Outcome of the Adverse Event.
Description: Adverse events were assessed at each visit through month 7 of the study. No subject discontinued valganciclovir therapy due to permanent discontinuation of valganciclovir therapy or lead to irreversible outcome of any adverse event.
Time Frame: baseline through 7 months
Measure: Number; unit: participants
Groups:
- Valganciclovir: 24 Wks Valganciclovir: Six months of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks Placebo | Valganciclovir: 24 Wks Valganciclovir
Number analyzed (Participants) | 49 | 47
participants
  Permanent discontinuation of study drug | 0 | 0
  Irreversible outcome from use of study drug | 0 | 0

3. Secondary Outcome: Change in Best Ear Hearing Assessments at 12 Months.
Description: Hearing assessment was evaluated by an independent audiologist. At baseline, a brainstem evoked response (BSER) assessment and autoacoustic emissions (OAEs) hearing assessments were obtained. At 12 months, BSER and /or Visual reinforcement audiometry (VRA) and OAEs were obtained. A single, independent study audiologist who was blinded to treatment assignment assessed the audiology test battery for each subject and assigned the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications were assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. Following this, the study audiologist assigned the "best ear" classification for the subject at that study visit; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification was mild hearing loss.
Time Frame: Between baseline and 12 months
Population: Only subjects randomized and subjects that had both baseline and 12 month hearing exams were analyzed for the primary endpoint. Some subjects failed to have the one or both of the two hearing exams (baseline and/or 12 months). There were 40 placebo subjects and 41 active drug subjects reported results for both time periods
Measure: Number; unit: participants
Groups:
- Valganciclovir: 24 Weeks of Valganciclovir: Six months of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Weeks of Valganciclovir
Number analyzed (Participants) | 40 | 41
participants
  Improved hearing | 2 | 2
  No change - normal hearing | 23 | 30
  No change - same degree of hearing loss | 10 | 6
  Worsening hearing | 5 | 3

4. Secondary Outcome: Change in Best Ear Hearing Assessments at 24 Months.
Description: Hearing assessment was evaluated by an independent audiologist. At baseline, a brainstem evoked response (BSER) assessment and autoacoustic emissions (OAEs) hearing assessments were obtained. At 24 months, BSER and /or Visual reinforcement audiometry (VRA) and OAEs were obtained. A single, independent study audiologist who was blinded to treatment assignment assessed the audiology test battery for each subject and assigned the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications were assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. Following this, the study audiologist assigned the "best ear" classification for the subject at that study visit; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification was mild hearing loss.
Time Frame: Between baseline and 24 months
Population: Only subjects randomized and subjects that had both baseline and 24 month hearing exams were analyzed for the primary endpoint. Some subjects failed to have the one or both of the two hearing exams (baseline and/or 24 months). There were 31 placebo subjects and 37 active drug subjects reported results for both time periods
Measure: Number; unit: participants
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 31 | 37
participants
  Improved hearing | 2 | 2
  No change - normal hearing | 20 | 30
  No change - same degree of hearing loss | 7 | 2
  Worsening hearing | 2 | 3

5. Secondary Outcome: Number of Ears With Improvement or Protected Hearing in Hearing Assessments Over Left and Right Ears at 6 Months.(Based on 84 Ears From 43 Placebo Subjects and 82 Ears From 43 Valganciclovir Subjects)
Description: as for outcome 1
Time Frame: Between baseline and 6 months
Population: as for outcome 1
Measure: Number; unit: ears
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 43 | 43
ears
  Improved or protected hearing | 46 | 52
  Same hearing loss or deterioration | 38 | 30

6. Secondary Outcome: Number of Ears With Improvement or Protected Hearing in Hearing Assessments Over Left and Right Ears at 12 Months.(Based on 77 Ears From 40 Placebo Subjects and 79 Ears From 41 Valganciclovir Subjects)
Description: as for outcome 3
Time Frame: Between baseline and 12 months
Population: Only subjects that were randomized and had baseline and 12 month hearing exams were analyzed.
Measure: Number; unit: ears
Groups:
- Placebo: Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
- Valganciclovir: Six months of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 40 | 41
ears
  Improved or protected hearing | 44 | 58
  Same hearing loss or worsening | 33 | 21

7. Secondary Outcome: Number of Ears With Improvement or Protected Hearing Assessments Over Left and Right Ears at 24 Months.(Based on 58 Ears From 31 Placebo Subjects and 70 Ears From 37 Valganciclovir Subjects)
Description: as for outcome 4
Time Frame: Between baseline and 24 months
Population: as for outcome 4
Measure: Number; unit: ears
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 31 | 37
ears
  Improved or protected | 37 | 54
  Same hearing loss or worsened hearing | 21 | 16

8. Secondary Outcome: Number of Ears With Hearing Deterioration Over Left and Right Ears at 6 Months.(Based on 84 Ears From 43 Placebo Subjects and 82 Ears From 43 Valganciclovir Subjects)
Description: as for outcome 1
Time Frame: Between baseline and 6 months
Population: as for outcome 1
Measure: Number; unit: ears
Groups:
- Placebo: 6 Wks of Vlaganciclovir Followed by 18 Wks of Placebo: Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
Arm/Group | Placebo: 6 Wks of Vlaganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 43 | 43
ears
  No worsening of hearing | 75 | 71
  Worsening hearing | 9 | 11

9. Secondary Outcome: Number of Ears With Hearing Deterioration Over Left and Right Ears at 12 Months.(Based on 77 Ears From 40 Placebo Subjects and 79 Ears From 41 Valganciclovir Subjects)
Description: as for outcome 3
Time Frame: Between baseline and 12 months
Population: as for outcome 3
Measure: Number; unit: ears
Groups:
- Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo: Six weeks of oral Valganciclovir followed by placebo to complete the six month time period.
  Placebo : 9 grams of powder which contains no Valganciclovir free base. The oral solution formulation comprises the following excipients: mannitol, lactose anhydrous, fumaric acid, sodium benzoate, saccharin sodium, flavor, and purified water.
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 40 | 41
ears
  No worsening of hearing | 67 | 73
  Worsening hearing | 10 | 6

10. Secondary Outcome: Number of Ears With Hearing Deterioration Over Left and Right Ears at 24 Months.(Based on 58 Ears From 31 Placebo Subjects and 70 Ears From 37 Valganciclovir Subjects)
Description: as for outcome 4
Time Frame: Between baseline and 24 months
Population: as for outcome 4
Measure: Number; unit: ears
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir
Number analyzed (Participants) | 31 | 37
ears
  No worsening of hearing | 53 | 62
  Worsening hearing | 5 | 8

11. Secondary Outcome: Neurological Impairment at 12 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Cognitive Composite Score).
Description: Cognitive Composite Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Composite Scores, the range of scores is between 40 (very poor cognitive skills) and 160 (excellent cognitive skills), with the average cogonitive skills score for a child (age adjusted) is 100 with standard deviation of 15.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam Cognitive Composite Score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 45 | 43
units on a scale | 76.5 (3.4) | 84.2 (3.0)

12. Secondary Outcome: Neurological Impairment at 12 Months of Age Utilizing the Bayley Scales of Infant and Toddler Development (Receptive Communication Scaled Score).
Description: Receptive Communication Scaled Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Scaled Scores, the range of scores is between 1 (very poor receptive communication skills) and 19 (excellent receptive communication skills), with the average receptive communication skills score for a child (age adjusted) is 10 with standard deviation of 3.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam Receptive Communications scorewere analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 43 | 41
units on a scale | 5.8 (0.5) | 6.8 (0.6)

13. Secondary Outcome: Neurological Impairment at 12 Months of Age Utilizing the Bayley Scales of Infant and Toddler Development (Expressive Communication Scaled Score).
Description: Expressive Communication Scaled Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Scaled Scores, the range of scores is between 1 (very poor expressive communication skills) and 19 (excellent expressive communication skills), with the average expressive communication skills score for a child (age adjusted) is 10 with standard deviation of 3.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam expressinve Communications scaled score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 44 | 41
units on a scale | 6.1 (0.5) | 7.3 (0.5)

14. Secondary Outcome: Neurological Impairment at 12 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Language Composite Score).
Description: Language Composite Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Composite Scores, the range of scores is between 40 (very poor language skills) and 160 (excellent language skills), with the average language skills score for a child (age adjusted) is 100 with standard deviation of 15.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam language composite score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir
Number analyzed (Participants) | 43 | 41
units on a scale | 74.8 (3.2) | 82.9 (2.9)

15. Secondary Outcome: Neurological Impairment at 12 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Fine Motor Scaled Score).
Description: Fine Motor Scaled Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Scaled Scores, the range of scores is between 1 (very poor fine motor skills) and 19 (excellent fine motor skills), with the average fine motor skills score for a child (age adjusted) is 10 with standard deviation of 3.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam fine motor score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir
Number analyzed (Participants) | 44 | 41
units on a scale | 5.5 (0.6) | 6.5 (0.6)

16. Secondary Outcome: Neurological Impairment at 12 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Gross Motor Scaled Score).
Description: Gross Motor Scaled Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Scaled Scores, the range of scores is between 1 (very poor gross motor skills) and 19 (excellent gross motor skills), with the average gross motor skills score for a child (age adjusted) is 10 with standard deviation of 3.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam gross motor score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 44 | 42
units on a scale | 4.9 (0.6) | 5.6 (0.5)

17. Secondary Outcome: Neurological Impairment at 12 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Motor Composite Score).
Description: Motor Composite Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Composite Scores, the range of scores is between 40 (very poor motor skills) and 160 (excellent motor skills), with the average motor skills score for a child (age adjusted) is 100 with standard deviation of 15.
Time Frame: 12 Months after enrollment
Population: only subjects that were randomized and had the 12 month Bayleys exam motor composite score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 44 | 42
units on a scale | 70.0 (3.7) | 76.5 (3.1)

18. Secondary Outcome: Neurological Impairment at 24 Months Utilizing the Bayley Scales of Infant and Toddler Development (Receptive Communication Scaled Score).
Description: as for outcome 12
Time Frame: 24 Months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam receptive communication scaled were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 41 | 41
units on a scale | 4.9 (0.5) | 6.4 (0.6)

19. Secondary Outcome: Neurological Impairment at 24 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Cognitive Composite Score).
Description: Cognitive Composite Score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring of the Composite Scores, the range of scores are between 40 (very poor cognitive skills) and 160 (excellent cognitive skills), with the average cognitive skills score for a child (age adjusted) is 100 with standard deviation of 15.
Time Frame: 24 months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam cognitive composite score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 41 | 42
units on a scale | 74.9 (2.8) | 79.6 (2.9)

20. Secondary Outcome: Neurological Impairment at 24 Months of Life, Utilizing the Bayley Scales of Infant and Toddler Development (Expressive Communication Scaled Score).
Description: as for outcome 13
Time Frame: 24 Months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam expressive communications scaled score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks Valganciclovir
Number analyzed (Participants) | 41 | 41
units on a scale | 5.3 (0.6) | 6.5 (0.5)

21. Secondary Outcome: Neurologic Impairment at 24 Months of Life Utilizing the Bayley Scales of Infant and Toddler Development (Language Composite Score).
Description: as for outcome 14
Time Frame: 24 Months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam language composite score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Valganciclovir: 24 Wks of Vlaganciclovir: Six months of oral Valganciclovir.
  Valganciclovir : Mono-valyl ester pro-drug of ganciclovir, oral solution, provided as a 12 grams of powder containing 5 grams of Valganciclovir free base. The oral solution formulation comprises the following excipients: Providone K30, fumaric acid, sodium benzoate, sodium saccharin, mannitol, flavor, and purified water.
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Vlaganciclovir
Number analyzed (Participants) | 41 | 41
units on a scale | 71.2 (3.3) | 79.5 (3.1)

22. Secondary Outcome: Neurological Impairment at 24 Months, Utilizing the Bayley Scales of Infant and Toddler Development (Fine Motor Scaled Score).
Description: as for outcome 15
Time Frame: 24 Months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam fine motor were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 40 | 42
units on a scale | 6.0 (0.7) | 6.9 (0.6)

23. Secondary Outcome: Neurological Impairment at 24 Months of Life, Utilizing the Bayley Scales of Infant and Toddler Development (Gross Motor Scaled Score).
Description: Gross motor scaled score for infants and toddlers was measured by use of the Bayley Scales of Infant and Toddler Development. For the Bayleys scoring is between 1 (very poor gross motor skills) and 19 (excellent gross motor skills), with the average gross motor skills score for a child (age adjusted) is 10 with standard deviation of 3.
Time Frame: 24 Months after enrollment.
Population: only subjects that were randomized and had the 24 month Bayleys exam gross motor score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 40 | 42
units on a scale | 4.9 (0.6) | 6.1 (0.5)

24. Secondary Outcome: Neurological Impairment at 24 Months of Life, Utilizing the Bayley Scales of Infant and Toddler Development (Motor Composite Score).
Description: as for outcome 17
Time Frame: 24 Months after enrollment
Population: only subjects that were randomized and had the 24 month Bayleys exam motor composite score were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo: 6 Wks of Valganciclovir Followed by 18 Wks of Placebo | Valganciclovir: 24 Wks of Valganciclovir
Number analyzed (Participants) | 40 | 41
units on a scale | 71.8 (3.7) | 80.1 (3.3)

ADVERSE EVENTS:
Time Frame: Adverse events were reported between baseline and 7 months
Description: There were three groups: 13 subjects who only received 6 weeks of open label valganciclovir (these 13 did not receive blinded study drug)); 47 subjects receive a full 24 weeks of valganciclovir and 49 subjects received 6 weeks of valganciclovir and 18 weeks of placebo.
Groups:
- Non Randomized: 6 weeks of open label valganciclovir only
- Active: 6 weeks of open labeled vanganciclovir followed by 4 1/2 months of blinded valganciclovir
- Placebo After 6 Weeks of Valganciclovir: 6 weeks of open labeled vanganciclovir followed by 4 1/2 months of blinded placebo
Arm/Group | Non Randomized | Active | Placebo After 6 Weeks of Valganciclovir
Serious Adverse Events (participants affected / at risk) | 1/13 | 11/47 | 19/49
Other Adverse Events (participants affected / at risk) | 3/13 | 45/47 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Randomized (N=13) | Active (N=47) | Placebo After 6 Weeks of Valganciclovir (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 8 (9)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomoting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis medial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Randomized (N=13) | Active (N=47) | Placebo After 6 Weeks of Valganciclovir (N=49)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (6) | 9 (13)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 11 (15) | 14 (33)
Neutropenia Neonatal (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 4 (4) | 4 (5)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Eye movement disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photalgia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 3 (3)
Swollen tear duct (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 13 (23)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 5 (6) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (6) | 10 (11)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3)
Infantile spitting up (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 9 (14) | 6 (12)
Developmental delay (General disorders) | 0 (0) | 2 (2) | 2 (2)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fever neonatal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 3 (4)
Irritability postvaccinal (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 8 (10)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (3) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
Candida nappy rash (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 5 (5) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 7 (9) | 6 (6)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 11 (15) | 12 (23)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis media bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Recurring skin boils (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 15 (24) | 14 (19)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 3 (5) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Bacteria stool identified (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 2 (4) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 2 (4) | 2 (2)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin abnormal (Investigations) | 0 (0) | 1 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Head lag (Investigations) | 0 (0) | 0 (0) | 3 (3)
Liver function test abnormal (Investigations) | 1 (1) | 6 (6) | 4 (7)
Neutrophil count abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 2 (2) | 3 (3)
Stool analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Crying (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4)
Infantile spasms (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (2) | 3 (3)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Reflexes abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep phase rhythm disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 6 (8)
Nasopharyngeal reflux (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (11) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7) | 11 (13)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Circumcision (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1)
Oxygen supplementation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days